CLINICAL TRIAL: NCT02010320
Title: Prospective Testing of Pharmacokinetic Population Models for Dosing of Transplanted Patients
Brief Title: Computer Guided Doing of Tacrolimus in Renal Transplantation
Acronym: OPTIMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Collaborators: Rikshospitalet University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMAL-13
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Renal Transplantation
Keywords: population model; pharmacokinetic; tacrolimus; therapeutic drug monitoring; individualized dosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer dosed (Experimental): Patients for which the computer model will calculate the individual doses
  Interventions: Other: Computer dosing
- Control (Active Comparator): Patients which will get their tacrolimus doses determined by experience transplant physicians
  Interventions: Other: Standard dose determination

INTERVENTIONS:
Other: Computer dosing — Pharmacokinetic population model for individual dose estimations of tacrolimus based on concentrations measurements and inclusion of relevant covariates
  Arms: Computer dosed
Other: Standard dose determination — Tacrolimus dose determination according to trough concentrations and standard TDM at the clinic
  Arms: Control

SUMMARY:
Dosing of tacrolimus is challenging due to the large inter-individual variation in its pharmacokinetics. The investigators have developed a pharmacokinetics population model that can be used to estimate individual doses of tacrolimus in renal transplant recipients. The model will be prospective tested in a randomized clinical trial.

The hypothesis is that the computer model is superior to experienced transplant physicians in reaching and keeping the patients in the target range of tacrolimus.

DETAILED DESCRIPTION:
Patients will be randomized to either computer or standard dosing strategies at time of transplantation or as early after transplantation as possible in case of deceased donor transplants.

For patients in the computer arm the model will calculate the dose with the highest probability to reach the specified concentration target.

For all concentrations a predictive error will be calculated and this will be the primary endpoint that the statistics will be calculated on.

All patients will be followed for between 8 to 12 weeks post-transplant, according to center praxis.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant recipients using tacrolimus as part of their immunosuppression
* above 18 years
* signed informed consent

Exclusion Criteria:

* no specific

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Predictive error (Cpred-Cobs) | 8 to 12 weeks
  Predictive error will be calculated as the computer predicted concentration minus the measured concentration over the first 8 to 12 weeks post-transplant in the computer group. The calculations will be binned into weekly assessments.
Reaching the target concentration | 8 to 12 weeks post-transplant
  In each arm the deviation of the observed concentration front he preset target concentration will be calculated for each measured concentration. The deviations will be compared between the two arms.

OTHER OUTCOMES:
Influence of CYP3A5 genotyping | 8 to 12 weeks post-transplant
  The model will be run without any information about patients CYP3A5 genotype as this is not clinical praxis at our center yet. All patients will however be genotyped after the study and a model including this covariate will be used to recalculate the data and see if this model is superior to the simple model, primary by comparing predictive errors in the computer arm.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, PhD, Study Chair — OUS-Rikshospitalet and University of Oslo
Locations (1):
- Olso university hospital - Rikshospitalet, Oslo, Norway

REFERENCES:
- [Derived] Storset E, Asberg A, Skauby M, Neely M, Bergan S, Bremer S, Midtvedt K. Improved Tacrolimus Target Concentration Achievement Using Computerized Dosing in Renal Transplant Recipients--A Prospective, Randomized Study. Transplantation. 2015 Oct;99(10):2158-66. doi: 10.1097/TP.0000000000000708. PMID 25886918